CLINICAL TRIAL: NCT00005383
Title: Anger and Cardiovascular Risk in Urban Youth
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4288; R01HL052080 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity

SUMMARY:
To examine anger and cardiovascular disease risk in urban youth. The project studied patterns of hemodynamic responses to social and nonsocial stressors, ambulatory blood pressure (BP), fasting insulin, fasting glucose, lipid profiles, and central obesity in adolescents from a wide range of socioeconomic status (SES) backgrounds.

DETAILED DESCRIPTION:
BACKGROUND:

Urban adolescents at high risk for cardiovascular disease (CVD) exhibit a pattern of hemodynamic responses that: (a) is evoked by social encounters that arouse anger, defensiveness, and distrust; (b) appears related to increased insulin resistance; (c) is more pronounced in males and African Americans; and (d) may constitute a pathway via which chronic exposure to stressful social environments increases CVD risk.

DESIGN NARRATIVE:

There were four studies. Study 1 in the first two years measured hemodynamics in 200 subjects to test the hypothesis that hostile distrust was associated with increased total peripheral resistance (TPR) response to social challenge, and that adolescents exhibiting this response pattern had elevated levels of ambulatory BP, fasting insulin, glucose, blood lipids, and central obesity. Study 2 followed 200 subjects for four years to determine if defensive hostility and distrust were related to tracking at higher levels of BP (measured every 6 months), and insulin/ glucose/ cholesterol (measured once per year). Study 3 in years 3 and 4 evaluated the influence of race on the cross-situational consistency of hostile distrust/BP by measuring the latter responses in 200 adolescents during structured encounters with a friend of the same race and sex, an unfamiliar same-race peer, and an unfamiliar other-race peer (black or white). Study 4 evaluated video and audiotape recordings from Studies 1 and 3 to test the hypothesis that distrustful individuals expressed more hostile affect in encounters with others, elicited more negative treatment, were perceived as hostile regardless of observer race or gender, and thus experienced chronic, health-damaging interpersonal stress. Study 4 data were used to examine the possibility that hostile distrust is related to exposure to crime, poverty, and racial discrimination.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-01; Study Completion 1999-12 (Actual)

REFERENCES:
- [Background] Ewart CK, Jorgensen RS, Kolodner KB. Sociotropic cognition moderates blood pressure response to interpersonal stress in high-risk adolescent girls. Int J Psychophysiol. 1998 Mar;28(2):131-42. doi: 10.1016/s0167-8760(97)00091-3. PMID 9545651
- [Background] Ewart CK, Suchday S. Discovering how urban poverty and violence affect health: development and validation of a Neighborhood Stress Index. Health Psychol. 2002 May;21(3):254-62. doi: 10.1037//0278-6133.21.3.254. PMID 12027031